CLINICAL TRIAL: NCT06094673
Title: The Relationship Between Systemic Immune Inflammation Index and Disease Activity in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH4
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; complete blood count; inflammation
MeSH Terms: conditions — Spondylitis, Ankylosing; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In this study, the aim was to investigate the relationship between SII and other laboratory parameters with disease activity in AS patients and to discuss its usability in the follow-up and treatment process.

DETAILED DESCRIPTION:
This study aimed to investigate the relationship between the systemic immune inflammation index (SII), platelet-to-lymphocyte ratio (PLR), neutrophil-to-lymphocyte ratio (NLR), and disease activity and functional status in patients with ankylosing spondylitis (AS). A cross-sectional clinical study was conducted, and a total of 90 patients diagnosed with AS according to the Modified New York Criteria, aged between 18 and 65, who presented to our outpatient clinics were included in the study. Demographic data, disease duration, age at symptom onset, and laboratory parameters, including platelet, neutrophil, basophil, eosinophil, lymphocyte counts, mean platelet volume (MPV), red blood cell distribution width (RDW), C-reactive protein (CRP), and erythrocyte sedimentation rate (ESR), were recorded. NLR and PLR values were calculated. The Systemic Immune Inflammation Index (SII) was calculated by dividing the product of neutrophil and platelet counts by the lymphocyte count. We investigated all of these parameters and disease activity scores. Disease activity was assessed with the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), spinal mobility with the Bath Ankylosing Spondylitis Metrology Index (BASMI), and functional status with the Bath Ankylosing Spondylitis Functional Index (BASFI). In addition, during the routine follow-ups of patients, requested blood tests were examined, and platelet, neutrophil, basophil, eosinophil, lymphocyte counts, mean platelet volume (MPV), RDW (red blood distribution width), CRP, and ESR values will be recorded. Neutrophil-lymphocyte ratio (NLR), platelet-lymphocyte ratio (PLR), and systemic immune inflammation index (SII) were calculated

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 65 who have been diagnosed with Ankylosing Spondylitis according to the Modified New York Criteria, have applied to the Istanbul Physical Medicine and Rehabilitation Training and Research Hospital outpatient clinic on the specified dates, meet the exclusion criteria, and have complete blood count, CRP, and ESR values in their hospital records.

Exclusion Criteria:

* Presence of acute or chronic infection

  * Presence of autoimmune diseases other than Ankylosing Spondylitis
  * Pregnancy
  * Diabetes
  * Chronic kidney disease
  * Chronic liver disease
  * Malignancy
  * Cardiovascular disease
  * Hematological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who have been diagnosed with Ankylosing Spondylitis according to the Modified New York Criteria
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
The Systemic Immune Inflammation Index (SII) | through study completion, an average of 1 month
  The Systemic Immune Inflammation Index (SII) was calculated by dividing the product of neutrophil and platelet counts by the lymphocyte count.
Neutrophil-to-lymphocyte ratio (NLR) | through study completion, an average of 1 month
  NLR is a ratio between the absolute neutrophil count and absolute lymphocyte count.
Platelet to-lymphocyte ratio (PLR) | through study completion, an average of 1 month
  PLR is a ratio between the absolute platelet count and absolute lymphocyte count.
Mean platelet volume (MPV) | through study completion, an average of 1 month
  MPV blood test measures the average size of patient's platelets
Red blood cell distribution width (RDW) | through study completion, an average of 1 month
  A red cell distribution width (RDW) test measures the differences in the volume and size of the red blood cells (erythrocytes).

SECONDARY OUTCOMES:
C-reactive protein | through study completion, an average of 1 month
  C-reactive protein (CRP) is a protein made by the liver. The level of CRP increases when there's inflammation in the body.
Erythrocyte sedimentation rate | through study completion, an average of 1 month
  The erythrocyte sedimentation rate (sedimentation rate, sed rate, or ESR for short) is a commonly performed hematology test that may indicate and monitor an increase in inflammatory activity within the body caused by one or more conditions such as autoimmune disease, infections, or tumors
The Bath Ankylosing Spondylitis Disease Activity Index | through study completion, an average of 1 month
  The index indicates that disease activity of AS patients. Higher scores indicate that higher activity
The Bath Ankylosing Spondylitis Functional Index | through study completion, an average of 1 month
  The index helps to evaluate disease activity of AS patients. High scores indicate that worse functional status.
The Bath Ankylosing Spondylitis Metrology Index | through study completion, an average of 1 month
  The index helps to evaluate spinal mobility of AS patients. Higher scores indicate more limited mobility.
Ankylosing Spondylitis Disease Activity Score with erythrocyte sedimentation rate | through study completion, an average of 1 month
  it helps to evaluate disease activity of AS patients by used to esr
Ankylosing Spondylitis Disease Activity Score with c-reactive protein | through study completion, an average of 1 month
  it helps to evaluate disease activity of AS patients by used to crp

CONTACTS AND LOCATIONS:
Overall Officials: Nur Kesiktas, MD, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Therapy and Rehabilitation Research and Training Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu J, Yan L, Chai K. Systemic immune-inflammation index is associated with disease activity in patients with ankylosing spondylitis. J Clin Lab Anal. 2021 Sep;35(9):e23964. doi: 10.1002/jcla.23964. Epub 2021 Aug 21. PMID 34418163
- [Result] Liang T, Chen J, Xu G, Zhang Z, Xue J, Zeng H, Jiang J, Chen T, Qin Z, Li H, Ye Z, Nie Y, Zhan X, Liu C. Platelet-to-Lymphocyte Ratio as an Independent Factor Was Associated With the Severity of Ankylosing Spondylitis. Front Immunol. 2021 Nov 5;12:760214. doi: 10.3389/fimmu.2021.760214. eCollection 2021. PMID 34804047
- [Result] Choe JY, Lee CU, Kim SK. Association between Novel Hematological Indices and Measures of Disease Activity in Patients with Rheumatoid Arthritis. Medicina (Kaunas). 2023 Jan 6;59(1):117. doi: 10.3390/medicina59010117. PMID 36676741
- [Result] Satis S. New Inflammatory Marker Associated with Disease Activity in Rheumatoid Arthritis: The Systemic Immune-Inflammation Index. Curr Health Sci J. 2021 Oct-Dec;47(4):553-557. doi: 10.12865/CHSJ.47.04.11. Epub 2021 Dec 31. PMID 35444819
- [Result] Seng JJB, Kwan YH, Low LL, Thumboo J, Fong WSW. Role of neutrophil to lymphocyte ratio (NLR), platelet to lymphocyte ratio (PLR) and mean platelet volume (MPV) in assessing disease control in Asian patients with axial spondyloarthritis. Biomarkers. 2018 May-Jun;23(4):335-338. doi: 10.1080/1354750X.2018.1425916. Epub 2018 Jan 24. PMID 29307233